CLINICAL TRIAL: NCT02782273
Title: The Analgesic Effects of Morphine Versus Ketorolac in Renal Colic
Brief Title: Morphine Versus Ketorolac in Renal Colic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loredana Ghinea (Other)
Responsible Party: Sponsor-Investigator, Loredana Ghinea, Medical Doctor, Bucharest Emergency Hospital
Organization: Bucharest Emergency Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-4627
Record Dates: First submitted 2016-05-16; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Renal Colic
Keywords: ketorolac; pain relieve; morphine
MeSH Terms: conditions — Renal Colic | interventions — Ketorolac; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac (Active Comparator): The patients randomised to this arm they will receive 30 mg intravenous ketorolac.
  Interventions: Drug: Morphine
- Morphine (Active Comparator): The patients randomised to this arm they will receive 0,1 mg/kg intravenous morphine.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — The patients randomised to this arm they will receive 30 mg intravenous ketorolac.
  Arms: Morphine
Drug: Morphine — The patients randomised to this arm they will receive 0,1 mg/kg intravenous morphine.
  Arms: Ketorolac

SUMMARY:
The study is prospective, double blinded, randomised controlled and has the purpose to compare the analgesic effects of ketorolac or morphine intravenous in renal colic.

DETAILED DESCRIPTION:
The study will take place in the Emergency Department of the Clinical Emergency Hospital Bucharest and will compare the analgesic effects of ketorolac tromethamine against morphine in renal colic.

The patients will be randomised to receive either ketorolac 30 mg intravenous (diluted in 20 ml of 0,9% saline) or morphine 0,1 mg/kg weight intravenous. A scale of 1-10 will be used for measuring the pain, and the effects of the treatment will be evaluated at 15 minutes and 30 minutes from the administration of the drugs. After 30 minutes if there is no significant reduction of the pain a rescue therapy will be used : chlorhydrate drotaverine 40 mg, xilocaine 100 mg, both diluted in 100 ml saline and the other medication not used from the study (morphine or ketorolac tromethamine).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of renal colic
* grade 5 pain on a 1-10 visual pain scale

Exclusion Criteria:

* contraindications of ketorolac or opioids
* pregnancy
* allergies to ketorolac or opioids
* refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Reducing the grade of pain | 15 minutes, 30 minutes
  To see the reducing of the pain on a scale 1-10 at two time points

SECONDARY OUTCOMES:
Time of staying in emergency department | 30 minutes, 1 hour, 2 hours
The necessity of urology consult - interventional measures | 7 days
  The patients will be called after 7 days to see if they needed urology consult and urological intervention
The cost of each treatment | 1 hour
  To evaluate the costs of treatment of each type of drug and/or rescue therapy
The necessity to use rescue therapy - pain > 5 grade | 30 minutes
  30 minutes from presentation in the ED - if the pain is still > 5 on a 1-10 scale
Side effects of each treatment | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dan Marinescu, MD, Principal Investigator — Clinical Emergency Hospital Bucharest

IPD SHARING:
Plan to Share IPD: Undecided